CLINICAL TRIAL: NCT01697176
Title: A 1-year Prospective, Multicenter, Non-Randomized, Observational, Study to Evaluate Optimal Improvement of Vein Graft Patency Long Term by the Implementation of Novel Endoscopic Harvesting Techniques
Brief Title: Optimal Improvement of Vein Graft Patency Long Term by the Implementation Of Novel Endoscopic Harvesting Techniques
Acronym: OPTION
Status: Completed | Type: Observational
Sponsor: Cardiopulmonary Research Science and Technology Institute (Other)
Collaborators: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTION
Record Dates: First submitted 2012-02-17; First posted 2012-10-02 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study of lone Coronary Artery Bypass Grafting procedures with endoscopic vein graft harvesting using best harvesting practices.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational study of 100 patients who will undergo routine coronary artery bypass grafting. Eligible candidates will undergo lone Coronary Artery Bypass Graft (CABG) procedures with endoscopic vein harvesting using best harvesting practices, defined as: systemic heparinization prior to vein manipulation, standardization of vein graft harvesting techniques, pressure limiting syringe and 3 month use of dual anti-platelet therapy. Patients will undergo a CT angiography at 30 days and 12 months to assess vein graft patency.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and able to provide consent
* Eligible for endoscopic vein harvesting
* Minimum of two non sequential vein grafts
* Willing to comply with requirements of protocol

Exclusion Criteria:

* Previous CABG
* Previous or concomitant valve surgery
* Any other concomitant cardiac procedure other than surgical ablation or incidental PFO repair
* Intolerance to Iodine or IV contrast that cannot be controlled with pre-medication
* Renal insufficiency with GFR measurement ≤ 40, unless dialysis dependent
* Abnormal platelet level defined as Plt Count >400,000
* Abnormal platelet function (hypercoagulable state) as evidenced by TEG testing
* Allergy to or presence of a condition that the investigator feels may prevent safe administration of ASA or Plavix post-operatively.
* Patient has a co-morbid condition that in the opinion of the investigator poses undue risk for successful endovascular harvesting of the vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Isolated CABG
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Optimal Improvement of Vein Graft Patency Long Term by the Implementation of Novel Endoscopic Harvesting Techniques | 12 months
  To demonstrate improved vein graft patency rates at 12 months for endoscopically harvest saphenous vein grafts by employment of modifications to existing techniques in vein graft handling during harvests. Vein graft patency will be measured at 30 days post CABG and at one year post CABG as evaluated by cardiac CT angiography or cardiac catheterization.

SECONDARY OUTCOMES:
OPTION | 12 months
  To develop a standardized approach for harvesting, handling and preparing vein grafts in the endoscopic approach. By capturing the following:
  1. Incidence of vein graft failure at the time of initial CABG as evaluated by transit time graft flow measurements
  2. Incidence of vein graft failure at post-operative day 30 as evaluated by cardiac CT angiography or cardiac catheterization
  3. Incidence of vein graft failure at each interval (30 day and 12 month) as categorized by:
     1. Harvested vessel
     2. vein graft destinations
     3. vein graft quality

CONTACTS AND LOCATIONS:
Overall Officials: David Moore, MD, Principal Investigator — The Heart Hospital Baylor Plano; Michael J Mack, MD, Principal Investigator — Cardiopulmonary Research Science and Technology Institute
Locations (2):
- United States (2):
  - CRSTI/Medical City Dallas, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas